CLINICAL TRIAL: NCT00580268
Title: Bipolar Disorder in Pregnancy and the Postpartum Period: Predictors of Morbidity
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Viguera, Adele, MD, Center for Women's Mental Health, Massachusetts General Hospital
Other Study IDs: 2005P001167; R01MH071762 (NIH); NCT00320645 (obsolete NCT alias)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Bipolar Disorder; Psychiatric Morbidity; Neonatal Outcome
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, urine, whole blood, saliva, amniotic fluid, breast milk
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- H: Pregnant women with bipolar disorder

SUMMARY:
The purpose of this study is to examine risk factors for relapse of bipolar disorder during pregnancy and the postpartum period. The main goal of this study is to find the risks that may make it more likely for a woman with bipolar disorder to experience a depressive, manic, or hypomanic episode during her pregnancy and the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

1. medically healthy adult women (ages 18-45) fulfilling DSM-IV criteria for bipolar disorder of any type (1 or 2) who are currently pregnant within 14 weeks gestation dated by last menstrual period;
2. euthymic at the time of conception;
3. able to give informed consent and comply with study procedures;
4. have a treating psychiatrist, physician or mental health clinician. Gravid women between the ages of 18 and 45

Exclusion Criteria:

1. active suicidality or homicidality;
2. active substance use disorder with 6 months prior to enrollment, or
3. positive urine drug screen at enrollment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: psychiatrists, referring obstetricians, community-based health centers, triage, and women who have previously given written permission to be contacted about research studies within the MGH Perinatal and Reproductive Psychiatry Program
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2005-08; Primary Completion 2010-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
psychiatric morbidity | 15 months

SECONDARY OUTCOMES:
obstetrical outcomes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adele C Viguera, MD, Principal Investigator — MGH
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Massachusetts Geral Hospital, Boston, Massachusetts

REFERENCES:
- See also: MGH Center for Women's Mental Health — http://www.womensmentalhealth.org